CLINICAL TRIAL: NCT03343509
Title: A Prospective, Multicentre, Double-Blinded Randomised Controlled Trial Comparing Topical Versus Oral Metronidazole in Reducing Post-Operative Pain Following Excisional Haemorrhoidectomy
Brief Title: Topical Versus Oral Metronidazole Following Excisional Haemorrhoidectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, MBChB, MD (Thesis), EdD, FACS, FRACS, Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MetHaemorrhoid
Record Dates: First submitted 2017-11-05; First posted 2017-11-17 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Hemorrhoids; Postoperative Pain
Keywords: Hemorrhoidectomy; Metronidazole; Postoperative analgesia
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A - Oral (Experimental): Oral metronidazole 400mg 3 times a day for 7 days Placebo ointment applied 3 time times a day for 7 days to affected region
  Interventions: Drug: Metronidazole Oral; Drug: Placebo Ointment
- Group B - Topical (Experimental): Topical metronidazole ointment 10% 3 times a day for 7 days Oral placebo tablets 3 times a day for 7 days
  Interventions: Drug: Metronidazole Ointment; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Metronidazole Oral — Oral Metronidazole
  Arms: Group A - Oral
Drug: Metronidazole Ointment — Metronidazole Ointment
  Arms: Group B - Topical
Drug: Placebo Oral Tablet — Placebo Tablet
  Arms: Group B - Topical
Drug: Placebo Ointment — Placebo Ointment
  Arms: Group A - Oral

SUMMARY:
This study aims to determine if topical metronidazole reduces pain more than oral metronidazole following excisional haemorrhoidectomy. The trial will be a multi-centered, patient and investigator blinded superiority trial with two parallel groups and a primary outcome of pain scores during 14 days after surgery.

Group A will receive oral metronidazole and placebo cream. Group B will receive placebo tablets and topical metronidazole cream.

DETAILED DESCRIPTION:
The pathogenesis of post-operative excisional haemorrhoidectomy pain is multi-factorial with secondary bacterial colonisation, inflammation and anal sphincter spasm/hypertonicity all purposed to play a role. Several pharmacological agents have been introduced in the last two decades targeting specific parts of the hypothesized pathway of pain pathogenesis showing promising improvements.

Metronidazole is part of the nitroimidazole class of antibiotics and primarily affects anaerobic bacteria and protozoa and traditionally has been used in surgical prophylaxis and treating anaerobic infections. It has been postulated to decrease pain following EH via two mechanisms; first by decreasing secondary bacterial colonisation and hence reducing post-operative inflammation; and second via a hitherto poorly understood direct anti-inflammatory response. The oral route has been initially investigated but topical administration has more recently been mooted for analgesia and theoretically reduces the unpleasant systemic side effects of oral administration. Our research group has recently completed a systematic review of both oral and topical administration of metronidazole. This review showed benefit in reducing postoperative haemorrhoidectomy pain from both routes of administration but this far there has been no comparison of the two routes.

Metronidazole has been proposed to have both anti-bacterial and pleiotropic anti-inflammatory properties but its precise mechanism of action is unknown. The increased understanding of this novel use of an agent with a known pharmacological profile will generally broaden our use of a simple, cheap and widespread agent. The investigators hope research into this drug will enable its use beyond that of haemorrhoidectomies, with possible pleiotropic applications into other similar operations.

Given the high prevalence of haemorrhoids in a vital segment of New Zealand's population, this research will contribute to improved outcomes for affected patients. Decreasing the significant post-operative pain will improve the quality of life for New Zealanders as well as affected populations worldwide. Socially and financially, it will enable earlier return to normal activity and reduce the burden on visits and readmissions to primary and secondary care, respectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing excisional haemorrhoidectomy

Exclusion Criteria:

* < 16 years of age
* Have a simultaneous operation other than excisional haemorrhoidectomy
* History of chronic pain
* Previous allergy/adverse reaction to metronidazole
* Patients unable to consent or complete data questionnaires due to cognitive impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Daily Post-Operative Pain | Day 7
  Daily Post-Operative Pain Measured on Visual Analogue Scale (0 to 10)

SECONDARY OUTCOMES:
Total Analgesia Use | Day 7
  Measured in Morphine Equivalent Doses
Complication Rates | Day 30
  Short term complication rates including adverse reactions, bleeding, paraesthesiae, urinary retention, readmission
Return to Normal Activity | Day 30 (Followed up until returned back to normal)
  Time to return back to normal activity
Return of Bowel Function | Day 7
  Time for first bowel motion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB, Principal Investigator — The University of Auckland
Locations (2):
- New Zealand (2):
  - Manukau SuperClinic, Counties Manukau District Health Board, Auckland
  - Ormiston Hospital, Auckland

IPD SHARING:
Plan to Share IPD: No
Not to be shared